CLINICAL TRIAL: NCT00240539
Title: Long-term Follow-Up Studies at Years 16-20, to Evaluate the Persistence of Immune Response of GSK Biologicals' Hepatitis B Vaccine in Newborns of HBeAg+ and HBsAg+ Mothers in Comparison With a Historical Control Group
Brief Title: Long Term Follow-Up Study 16-20 Years After Hepatitis B Vaccination in Newborns of Mothers Who Were Seropositive for Hepatitis B Envelope Antigen (HBeAg) & Hepatitis B Surface Antigen (HBsAg)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 100449
Record Dates: First submitted 2005-10-13; First posted 2005-10-18 (Estimated); Results first posted 2009-11-17 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-10

CONDITIONS: Hepatitis B
Keywords: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Blood Specimen Collection

ARMS (4):
- HBsAg(+) & HBeAg(-) 4-dose Group (Experimental): Newborns of anti-hepatitis B surface antigen positive [HBsAg(+)] and hepatitis B envelope antigen negative [HBeAg(-)] mothers, who received 4 doses of Engerix™ in the primary study.
  Interventions: Procedure: Blood sampling
- HBsAg(+) & HBeAg(+) 4-dose Group (Experimental): Newborns of anti-hepatitis B surface antigen positive [HBsAg(+)] and hepatitis B envelope antigen positive [HBeAg(+)] mothers, who received 4 doses of Engerix™ in the primary study.
  Interventions: Procedure: Blood sampling
- HBsAg(+) & HBeAg(+) 5-dose Group (Experimental): Newborns of anti-hepatitis B surface antigen positive [HBsAg(+)] and hepatitis B envelope antigen positive [HBeAg(+)] mothers, who received 5 doses of Engerix™ in the primary study.
  Interventions: Procedure: Blood sampling
- HBsAg(-) & HBeAg(-) 4-dose Group (Experimental): Newborns of anti-hepatitis B surface antigen negative [HBsAg(-)] and hepatitis B envelope antigen negative [HBeAg(-)] mothers, who received 4 doses of Engerix™ in the primary study.
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — A blood sample will be taken yearly at each long-term follow-up time point (i.e. Year 16 through Year 20) after the first dose of Engerix-B™ vaccine.

SUMMARY:
This study is performed to evaluate the persistence of anti-hepatitis B surface antigen (HBs) antibodies up to 16, 17, 18, 19 and 20 years after administration of the first dose of the study vaccine, Engerix-B™. No new subjects will be recruited in this long-term follow-up study.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
The primary study was to evaluate the immunogenicity and protective efficacy of hepatitis B vaccine administered according to a 0, 1, 2, 12 month schedule in newborns of anti-hepatitis B envelope antigen positive (HBeAg+) and anti-hepatitis B surface antigen positive (HBsAg+) mothers. Results from the primary study have shown that the vaccine was immunogenic and protected neonates of HBeAg positive mothers against hepatitis B chronic carriage. The present study is carried out to evaluate the anti-HBs persistence and the prevalence and incidence of other hepatitis B markers (HBsAg, anti-hepatitis B core antigen {anti-HBc}, HBeAg, Alanine aminotransferase/Aspartate aminotransferase {ALT/AST}), and the clinical significance of the HBsAg and anti-HBc positive cases observed during the long-term from year 16-20. No vaccine will be administered during the long term follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who had participated in the primary study.
* Written informed consent obtained from the subject.

Ages: 16 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2003-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Poovorawan Y, Chongsrisawat V, Theamboonlers A, Srinivasa K, Hutagalung Y, Bock HL, Hoet B. Long-term benefit of hepatitis B vaccination among children in Thailand with transient hepatitis B virus infection who were born to hepatitis B surface antigen-positive mothers. J Infect Dis. 2009 Jul 1;200(1):33-8. doi: 10.1086/599331. PMID 19473096
- [Background] Poovorawan Y et al. Persistence of anti-HBs antibodies and immune memory 20-years after hepatitis B vaccination among children in Thailand. Abstract presented at the 9th International Congress of Tropical Pediatrics (ICTP). Bangkok, Thailand. 18-20 October 2011.
- [Derived] Poovorawan Y, Chongsrisawat V, Theamboonlers A, Crasta PD, Messier M, Hardt K. Long-term anti-HBs antibody persistence following infant vaccination against hepatitis B and evaluation of anamnestic response: a 20-year follow-up study in Thailand. Hum Vaccin Immunother. 2013 Aug;9(8):1679-84. doi: 10.4161/hv.24844. Epub 2013 May 31. PMID 23732904
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 100449 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 100449 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 100449 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 100449 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 100449 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant Flow and Baseline measures are given for the year 20 time point in order to account for all subjects participating in this long-term follow-up study.
  Note that not all subjects returned and participated in each of the intermediate follow-up time points.
Groups:
- HBsAg(+) & HBeAg(-) 4-dose Group: Newborns of HBsAg(+) and HBeAg negative [HBeAg(-)] mothers, who received 4 doses of Engerix™ in the primary study.
- HBsAg(+) & HBeAg(+) 4-dose Group: Newborns of HBsAg(+) and HBeAg(+) mothers, who received 4 doses of Engerix™ in the primary study.
- HBsAg(-) & HBeAg(-) 4-dose Group: Newborns of HBsAg(-) and HBeAg(-) mothers, who received 4 doses of Engerix™ in the primary study.
Period: Overall Study
Arm/Group | HBsAg(+) & HBeAg(+) 5-dose Group | HBsAg(+) & HBeAg(-) 4-dose Group | HBsAg(+) & HBeAg(+) 4-dose Group | HBsAg(-) & HBeAg(-) 4-dose Group
Started | 2 | 2 | 31 | 1
Completed | 2 | 2 | 31 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HBsAg(+) & HBeAg(+) 5-dose Group | HBsAg(+) & HBeAg(-) 4-dose Group | HBsAg(+) & HBeAg(+) 4-dose Group | HBsAg(-) & HBeAg(-) 4-dose Group | Total
Number analyzed (Participants) | 2 | 2 | 31 | 1 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 31 | 1 | 36
  >=65 years | 0 | 0 | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 2 | 2 | 18 | 1 | 23
  Male | 0 | 0 | 13 | 0 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Seropositive for Anti-hepatitis B Surface Antigen (Anti-HBs) Antibodies
Description: Seropositive subjects are subjects with anti-HBs antibody concentration ≥ 3.3 mIU/mL.
Time Frame: At Years 16, 17, 18, 19 and 20 after primary vaccination
Population: The analyses were performed on the Long-Term According to protocol (ATP) cohort for immunogenicity. Due to subjects being lost to follow up or eliminated from the ATP cohort for immunogenicity, no data from subjects in HBsAg(+) & HBeAg(-) 4-dose Group and HBsAg(-) & HBeAg(-) 4-dose Group were analyzed.
Measure: Number; unit: subjects
Arm/Group | HBsAg(+) & HBeAg(+) 5-dose Group | HBsAg(+) & HBeAg(-) 4-dose Group | HBsAg(+) & HBeAg(+) 4-dose Group | HBsAg(-) & HBeAg(-) 4-dose Group
Number analyzed (Participants) | 2 | 0 | 25 | 0
subjects
  Year 16 (n= 0, 25) | 0 [0 to 0] |  | 22 [22.7 to 86.7] |
  Year 17 (n= 2, 24) | 2 [0.2 to 765.3] |  | 21 [18.8 to 76.0] |
  Year 18 (n= 1, 22) | 1 [4.8 to 4.8] |  | 20 [18.9 to 65.7] |
  Year 19 (n= 2, 22) | 2 [0.0 to 2932.5] |  | 19 [14.8 to 59.5] |
  Year 20 (n= 2, 25) | 2 [4.0 to 14.9] |  | 23 [12.1 to 34.2] |

2. Primary Outcome: Number of Subjects Who Tested Positive for Markers of Infection With Hepatitis B Virus
Description: Tested markers were hepatitis B surface antigen (HBsAg), antibody to hepatitis B core antigen (anti-HBc), hepatitis B envelope antigen (HBeAg) and antibody to hepatitis B envelope antigen (anti-HBe).
Time Frame: At Years 16, 17, 18,19 and 20 after primary vaccination
Population: The analyses were performed on the ATP cohort for immunogenicity. Only subjects positive for HBsAg or anti-HBc markers were tested for HBeAg and anti-HBe markers for Year 17 to Year 20.
Measure: Number; unit: subjects
Arm/Group | HBsAg(+) & HBeAg(+) 5-dose Group | HBsAg(+) & HBeAg(-) 4-dose Group | HBsAg(+) & HBeAg(+) 4-dose Group | HBsAg(-) & HBeAg(-) 4-dose Group
Number analyzed (Participants) | 2 | 0 | 25 | 0
subjects
  HBsAg [Year 16] (n= 1, 25) | 0 |  | 0 |
  HBsAg [Year 17] (n= 2, 25) | 0 |  | 1 |
  HBsAg [Year 18] (n= 1, 22) | 0 |  | 0 |
  HBsAg [Year 19] (n= 1, 22) | 0 |  | 2 |
  HBsAg [Year 20] (n= 2, 25) | 0 |  | 2 |
  Anti-HBc [Year 16] (n= 1, 25) | 1 |  | 4 |
  Anti-HBc [Year 17] (n= 2, 25) | 1 |  | 3 |
  Anti-HBc [Year 18] (n= 1, 22) | 1 |  | 2 |
  Anti-HBc [Year 19] (n= 2, 22) | 1 |  | 2 |
  Anti-HBc [Year 20] (n= 2, 25) | 1 |  | 3 |
  HBeAg [Year 16] (n= 1, 23) | 0 |  | 0 |
  HBeAg [Year 17] (n= 1, 3) | 0 |  | 0 |
  HBeAg [Year 18] (n= 1, 2) | 0 |  | 0 |
  HBeAg [Year 19] (n= 1, 4) | 0 |  | 0 |
  HBeAg [Year 20] (n= 1, 5) | 0 |  | 0 |
  Anti-HBe [Year 16] (n= 1, 23) | 1 |  | 0 |
  Anti-HBe [Year 17] (n= 1, 4) | 1 |  | 1 |
  Anti-HBe [Year 18] (n= 1, 2) | 1 |  | 0 |
  Anti-HBe [Year 19] (n= 1, 4) | 0 |  | 0 |
  Anti-HBe [Year 20] (n= 1, 5) | 1 |  | 0 |

3. Primary Outcome: Number of Subjects With Chronic and With Clinical HBV Infection
Description: * Chronic HBV infection: HBsAg+ and anti-HBc+ at more than 2 consecutive time points.
  * Clinical HBV infection: Serologically confirmed, symptomatic HBV infection, and all HBV markers negative at consecutive time point.
Time Frame: From year 16 through to year 20
Measure: Number; unit: subjects
Arm/Group | HBsAg(+) & HBeAg(+) 5-dose Group | HBsAg(+) & HBeAg(-) 4-dose Group | HBsAg(+) & HBeAg(+) 4-dose Group | HBsAg(-) & HBeAg(-) 4-dose Group
Number analyzed (Participants) | 2 | 2 | 31 | 1
subjects
  Chronic HBV infection | 0 | 0 | 1 | 0
  Clinical HBV infection | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: No Adverse Event information was collected during this study
Arm/Group | HBsAg(+) & HBeAg(+) 5-dose Group | HBsAg(+) & HBeAg(-) 4-dose Group | HBsAg(+) & HBeAg(+) 4-dose Group | HBsAg(-) & HBeAg(-) 4-dose Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
No safety data were collected during this long-term follow-up study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.